CLINICAL TRIAL: NCT03444506
Title: A Single-Center, Double-Blind, Double-Dummy, Randomized, Parallel-Group, Comparative Environmental Exposure Chamber (EEC) Study to Evaluate Efficacy, Safety and Tolerability of Two Fixed Dose Combination (FDC) Products of Olopatadine Hydrochloride and Mometasone Furoate Nasal Spray as Compared to the FDC of Azelastine Hydrochloride and Fluticasone Propionate Nasal Spray, Olopatadine Nasal Spray, and Placebo in Patients With Seasonal Allergic Rhinitis.
Brief Title: Efficacy and Safety of Fixed Dose Combination (FDC) of Olopatadine Hydrochloride and Mometasone Furoate Nasal Spray (Molo; Also Referred as GSP 301) in the Treatment of Seasonal Allergic Rhinitis (SAR)
Acronym: GSP 301- PoC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glenmark Pharmaceuticals Ltd. India (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GPL/CT/2013/001/II
Record Dates: First submitted 2018-02-15; First posted 2018-02-23 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: SAR
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo nasal spray (Placebo Comparator): Placebo nasal spray - 2 sprays per nostril, BID
  Interventions: Drug: Placebo nasal spray
- Molo 1 (also referred as GSP 301-2 NS) (Experimental): Fixed Dose Combination of Molo nasal spray (olopatadine hydrochloride 665 mcg and mometasone furoate 25 mcg nasal spray) - 2 sprays per nostril, BID
  Interventions: Drug: Molo 1 (also referred as GSP 301-2 NS)
- Molo 2 (also referred as GSP 301-1 NS) (Experimental): Fixed Dose Combination of Molo nasal spray (olopatadine hydrochloride 665 mcg and mometasone furoate 50 mcg nasal spray) - 2 sprays per nostril, QD
  Interventions: Drug: Molo 2 (also referred as GSP 301-1 NS)
- DYMISTA nasal spray (Active Comparator): Fixed Dose Combination of azelastine hydrochloride 137 mcg and fluticasone propionate 50 mcg nasal spray - 1 spray per nostril, BID
  Interventions: Drug: DYMISTA nasal spray
- PATANASE nasal spray (Active Comparator): Olopatadine hydrochloride 665 mcg nasal spray - 2 sprays per nostril, BID
  Interventions: Drug: PATANASE nasal spray

INTERVENTIONS:
Drug: Molo 1 (also referred as GSP 301-2 NS)
  Arms: Molo 1 (also referred as GSP 301-2 NS)
Drug: Molo 2 (also referred as GSP 301-1 NS)
  Arms: Molo 2 (also referred as GSP 301-1 NS)
Drug: Placebo nasal spray
  Arms: Placebo nasal spray
Drug: DYMISTA nasal spray
  Arms: DYMISTA nasal spray
Drug: PATANASE nasal spray
  Arms: PATANASE nasal spray

SUMMARY:
A single-center, double-blind, placebo-controlled study of FDC olopatadine hydrochloride and mometasone furoate nasal spray (Molo; also referred as GSP 301) was conducted in subjects with seasonal allergic rhinitis. In this study, the efficacy and safety of two regimens (BID and QD) of the FDC (i.e. Molo 1 and Molo 2) were evaluated compared to placebo nasal spray, DYMISTA® and PATANASE®.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 to 65 years (inclusive) with a clinical history of seasonal allergic rhinitis (SAR) (for at least 2 years) and exhibiting a positive skin prick test

Exclusion Criteria:

* Pregnant or lactating women
* Patients with known hypersensitivity to any of the components of the formulation
* Patients with a history of seasonal asthma during ragweed season.
* Patient requiring chronic use of inhaled or systemic corticosteroids
* Patients with perennial rhinitis; non-allergic rhinitis; or ocular infection within 3 weeks before the screening
* Patients with history of acute or significant chronic sinusitis or chronic purulent post-nasal drip or Rhinitis Medicamentosa as determined by the Investigator.
* Patients with history of narrow-angle glaucoma, increased intraocular pressure, posterior subcapsular cataract, urinary retention, uncontrolled hypertension, severe Coronary Artery Disease, Ischemic Heart Disease, uncontrolled Diabetes Mellitus, Hyperthyroidism, Renal Impairment or Prostatic Hypertrophy, and those receiving MAO inhibitor therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-01-27 (Actual); Primary Completion 2014-02-28 (Actual); Study Completion 2014-02-28 (Actual)

PRIMARY OUTCOMES:
Change in mean post-treatment instantaneous Total Nasal Symptoms Score (iTNSS) for Molo 1 and Molo 2 compared with placebo from baseline to end of treatment | 15 days
  Instantaneous Total Nasal Symptom Score (iTNSS) is calculated as the sum of instantaneous scoring of the severity of four individual nasal symptoms (nasal congestion, rhinorrhea, nasal itching, sneezing). Subject responds on a 4-point severity scale with scores ranging from 0 (no signs/absent) to 3 (severe signs).

SECONDARY OUTCOMES:
Change in mean post-treatment iTNSS for Molo 1 and Molo 2 compared with reference products Dymista and Patanase | 15 days
  Instantaneous Total Nasal Symptom Score (iTNSS) is calculated as the sum of instantaneous scoring of the severity of four individual nasal symptoms (nasal congestion, rhinorrhea, nasal itching, sneezing). Subject responds on a 4-point severity scale with scores ranging from 0 (no signs/absent) to 3 (severe signs).
Change in mean post-treatment iTNSS for reference products Dymista and Patanase compared with placebo | 15 days
  Instantaneous Total Nasal Symptom Score (iTNSS) is calculated as the sum of instantaneous scoring of the severity of four individual nasal symptoms (nasal congestion, rhinorrhea, nasal itching, sneezing). Subject responds on a 4-point severity scale with scores ranging from 0 (no signs/absent) to 3 (severe signs).
Onset of action assessed by comparing change in iTNSS after the first dose | 15 days
Change from baseline in post-treatment instantaneous Total Symptoms Score (iTSS) (Molo 1 and Molo 2 versus Active Comparator) | 15 days
  Instantaneous Total Symptom Score (iTSS) is calculated as the sum of the four individual nasal symptom (nasal congestion, rhinorrhea, nasal itching, sneezing) scores and the three individual ocular symptom (ocular itching, tearing/watering eyes, and ocular redness) scores. Subject responds on a 4-point severity scale with scores ranging from 0 (no signs/absent) to 3 (severe signs).
Change from baseline in individual instantaneous Nasal Symptoms Scores (iNSS) (Molo 1 and Molo 2 versus Active Comparator) | 15 days
  Individual Instantaneous Nasal Symptoms Scores (iNSS) is calculated as the score of individual nasal symptoms (nasal congestion, rhinorrhea, nasal itching, sneezing). Subject responds on a 4-point severity scale with scores ranging from 0 (no signs/absent) to 3 (severe signs).
Change from baseline in instantaneous Total Ocular Symptom Score (iTOSS) (Molo 1 and Molo 2 versus Active Comparator) | 15 days
  Instantaneous Total Ocular Symptom Score (iTOSS) is calculated as the sum of the three individual ocular symptoms (ocular itching, tearing/watering eyes, and ocular redness). Subject responds on a 4-point severity scale with scores ranging from 0 (no signs/absent) to 3 (severe signs).
Change in mean post-treatment Environmental Exposure Chamber - Rhinoconjunctivitis Quality-of-Life Questionnaire (EEC-QoLQ) scores | 15 days
  The EEC-QoLQ has questions in three domains (non-nose/eye symptoms, practical problems and emotional) related to how much a subject was bothered with symptoms. Subject responds on a 7-point scale with score ranging from 0 (better outcome) to 6 (worse outcome).
Responses to a reflective Global Assessment of Tolerability and Acceptance Questionnaire (GATAQ) | 15 days
  Scale of 0 (very much acceptable) - 6 (not acceptable)

CONTACTS AND LOCATIONS:
Overall Officials: Sudeesh Tantry, PhD, Study Director — Glenmark Pharmaceuticals
Locations (1):
- Glenmark Investigational Site 1, Mississauga, Ontario, Canada

REFERENCES:
- [Derived] Patel P, Salapatek AM, Tantry SK. Effect of olopatadine-mometasone combination nasal spray on seasonal allergic rhinitis symptoms in an environmental exposure chamber study. Ann Allergy Asthma Immunol. 2019 Feb;122(2):160-166.e1. doi: 10.1016/j.anai.2018.10.011. Epub 2018 Oct 12. PMID 30321655